CLINICAL TRIAL: NCT01709383
Title: Can Enhancing Left Lateralization Using Transcranial Direct Current Stimulation Improve Recovery From Post-Stroke Aphasia?
Brief Title: Using Transcranial Direct Current Stimulation (tDCS) to Improve Post-Stroke Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DDCF 2012062
Record Dates: First submitted 2012-08-28; First posted 2012-10-18 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2016-10

CONDITIONS: Aphasia
Keywords: Aphasia; Stroke; Transcranial Direct Current Stimulation; Neuroplasticity
MeSH Terms: conditions — Aphasia; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Direct Current Stimulation (Active Comparator): TDCS was applied bilaterally, with the anodal electrode on the left temple and cathodal electrode on the right. TDCS was applied at the beginning of 60-minute speech-language treatment sessions for five days across a one-week period
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham Stimulation (Sham Comparator): Sham tDCS was applied at the beginning of 60-minute speech-language treatment sessions for five days across a one-week period.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — The tDCS treatments will be applied bilaterally, with the anodal electrode placed on the left temple and the cathodal electrode placed on the right temple. The tDCS will be applied at the beginning of 60-minute speech-language treatment sessions for five days across a one-week period.
  Arms: Transcranial Direct Current Stimulation
Device: Sham Stimulation — The sham tDCS will be applied at the beginning of 60-minute speech-language treatment sessions for five days across a one-week period.
  Arms: Sham Stimulation

SUMMARY:
This study tests whether weak electrical stimulation of the brain is effective in improving language or reading difficulties occurring after a brain injury or stroke.

DETAILED DESCRIPTION:
This study tests whether aphasia or alexia, language and reading disorders occurring after traumatic brain injury or stroke, can be improved using transcranial direct current stimulation (tDCS). tDCS is a non-invasive technique that applies a small amount of direct electrical current to the brain in order to temporarily alter brain processing. Adults with aphasia/alexia resulting from stroke or traumatic brain injury will undergo baseline behavioral testing of various language and cognitive functions. Subjects who are willing to undergo MRI evaluation will also be scanned. They will then receive five days of either real or sham tDCS with standardized speech-language therapy, under a double-blind randomized placebo-controlled design. Behavioral assessments, and MRIs for those participating in the MRI portion of the study, will be performed again at multiple time points after completing tDCS to assess for changes in these measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Aphasia due to left hemisphere stroke diagnosed by a physician or speech-language pathologist

Exclusion Criteria:

* Skull defect at or near the site of tDCS delivery
* History of a significant stroke or traumatic brain injury other than the event that caused the aphasia
* History of other brain conditions that could impact interpretation of results (such as multiple sclerosis, brain tumor, encephalitis, premorbid dementia)
* Presence of implanted electrical or metallic devices in the head or body (except titanium; e.g. cochlear implants, implanted shunts with metal parts, deep brain stimulators, pacemakers, defibrillators)
* Presence of ferrous metal in the head (e.g. shrapnel)
* History of psychiatric disease requiring hospitalization, electroconvulsive therapy, or ongoing medication use (other than common selective serotonin reuptake inhibitor antidepressants)
* Pregnancy
* Severe comprehension deficits

Additional Exclusion Criteria for the optional MRI portion of the study:

* Presence of metal in the body (except titanium)
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-12; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Turkeltaub, M.D., Ph.D., Principal Investigator — Georgetown University and MedStar National Rehabilitation Hospital
Locations (2):
- United States (2):
  - MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia
  - Georgetown University, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zaghi S, Acar M, Hultgren B, Boggio PS, Fregni F. Noninvasive brain stimulation with low-intensity electrical currents: putative mechanisms of action for direct and alternating current stimulation. Neuroscientist. 2010 Jun;16(3):285-307. doi: 10.1177/1073858409336227. Epub 2009 Dec 29. PMID 20040569
- [Result] Schlaug G, Marchina S, Wan CY. The use of non-invasive brain stimulation techniques to facilitate recovery from post-stroke aphasia. Neuropsychol Rev. 2011 Sep;21(3):288-301. doi: 10.1007/s11065-011-9181-y. Epub 2011 Aug 14. PMID 21842404
- [Result] Fridriksson J, Richardson JD, Baker JM, Rorden C. Transcranial direct current stimulation improves naming reaction time in fluent aphasia: a double-blind, sham-controlled study. Stroke. 2011 Mar;42(3):819-21. doi: 10.1161/STROKEAHA.110.600288. Epub 2011 Jan 13. PMID 21233468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusionary criteria were as follows: over 18; aphasia due to left hemisphere stroke; no other significant brain damage, neurological, or psychiatric disease; no skull defects near electrode sites; no implanted devices or ferrous metal in the body; not pregnant; comprehension sufficient to perform study tasks
Pre-assignment Details: Before randomization, potential subjects were tested on the Western Aphasia Battery -Revised (WAB-R) to determine a baseline score and to rule out severe comprehension deficits.
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Started | 24 | 14
Completed Treatment | 24 | 14
Completed Follow-ups | 23 | 14
Included in Analysis | 22 | 13
Completed | 23 | 14
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: People with aphasia due to left hemisphere stroke
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 24 | 14 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (10.8) | 59.8 (8.7) | 60.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 16 | 9 | 25
Region of Enrollment [Number; unit: participants]
  United States | 24 | 14 | 38

OUTCOME MEASURES:

1. Primary Outcome: Western Aphasia Battery - Revised: Naming and Word Finding Score
Description: This is a composite measure of verbal expression skills including tests of naming, verbal fluency, sentence completion, and responsive naming (one-word answers to basic questions). It is a subtest within the Western Aphasia Battery. The minimum score is 0 and maximum is 10, with 10 being the best outcome, and subscores are summed to determine the total score.
Time Frame: Change from baseline to one day after treatment
Population: People with aphasia due to left hemisphere stroke
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 22 | 13
scores on a scale | .30 (.64) | .48 (.74)
Statistical Analysis 1: Comparison: Transcranial Direct Current Stimulation vs Sham Stimulation; Test type: Superiority or Other; p = .57, Mixed Models Analysis

2. Secondary Outcome: Western Aphasia Battery - Revised: Spontaneous Speech, Repetition, Auditory Verbal Comprehension and Overall Aphasia Quotient
Description: The above subtests will reflect the following: a composite measure of information content in conversational speech and picture description (scored from 0 (no speech produced or only meaningless utterances) to 10 (no signs of aphasia)); a measure of word and sentence repetition (scored from 0 (unable to repeat any part of a single word) to 100 (perfect repetition of all words and up to a 10 word sentence)); a composite measure of yes/no questions, auditory word recognition, and following sequential commands (composite subscore is from 1 to 10, with 10 being the best outcome); and an overall aphasia severity score (composite score, or Aphasia Quotient, comprised of all the above measures plus the naming and word finding score used as the primary outcome measure. Quotient scores range from 0 to 100, with 100 indicating no aphasia is present).
Time Frame: Change from baseline to 1 day after treatment
Population: People with aphasia due to left hemisphere stroke
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 23 | 14
scores on a scale
  Spontaneous Speech Baseline | 7.6 (2.0) | 7.1 (2.8)
  Spontaneous Speech 1 day post-treatment | 7.8 (2.4) | 7.0 (2.9)
  Repetition Baseline | 5.5 (2.9) | 6.2 (2.9)
  Repetition 1 Day post-treatment | 5.8 (2.8) | 6.2 (3.1)
  Auditory Verbal Comprehension Baseline | 7.9 (1.3) | 8.0 (1.9)
  Auditory Verbal Comprehension 1 day post | 8.1 (1.4) | 7.8 (1.9)
  Aphasia Quotient Baseline | 66.2 (21.7) | 61.9 (28.6)
  Aphasia Quotient 1 Day post-treatment | 66.2 (21.7) | 65.1 (26.7)

3. Secondary Outcome: Philadelphia Naming Test (PNT)
Description: A test of picture naming using more common items than other picture naming tests, which reduces relationships between performance and premorbid education and socioeconomic status. There are 60 items on the test. A score of 0 means no pictures were named correctly. A score of 60 means all pictures were named correctly.
Time Frame: 1 day after treatment
Population: People with aphasia due to left hemisphere stroke
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 23 | 14
scores on a scale
  PNT Score Baseline | 31.3 (17.8) | 32.1 (23.5)
  PNT Score 1 Day Post-treatment | 34.1 (21.1) | 34.9 (3.1)
Statistical Analysis 1: Comparison: Transcranial Direct Current Stimulation vs Sham Stimulation; Test type: Superiority or Other; p = .64, Mixed Models Analysis

4. Secondary Outcome: Subjective Assessments Including: Communicative Effectiveness Index (CETI), Stroke and Aphasia Quality of Life Scale (SAQOL), and Stroke Aphasic Depression Questionnaire (SADQ)
Description: Questionnaires were given at baseline, 3 weeks and 3 months after treatment. The SADQ consists of 21 questions graded on a 0-3 scale with 3 indicating the highest depression symptoms and 0 indicating none. Therefore, means reported below are an average score between 0 and 3. The SAQOL includes 17 questions about functional physical limitations and 7 questions about functional communication limitations in daily life. Questions are rated on a 1-5 scale with a score of 1 indicating greater disability and 5 indicating none. Therefore, means reported below are an average score between 1 and 5. The CETI measures change in functional communication by asking caregivers to make a mark on a straight line with "as able as before the stroke" written on the right side of the line and "not at all as able" on the left. The 16 responses are then converted by measuring the location of the mark on the line. A score of 10 indicates "as able as before the stroke" and 0 indicates "not at all as able".
Time Frame: 3 weeks post-treatment
Population: People with aphasia due to left hemisphere stroke
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 18 | 10
scores on a scale
  SADQ Baseline | 1.2 (.2) | 1.58 (.4)
  SADQ 3 weeks post-treatment | 1.0 (.3) | 1.3 (.4)
  SAQOL Baseline | 2.7 (.7) | 2.6 (.7)
  SAQOL 3 weeks post-treatment | 2.9 (.8) | 2.7 (.9)
  CETI Baseline | 5.7 (1.7) | 6.8 (1.9)
  CETI 3 weeks post-treatment | 6.6 (2.0) | 6.4 (1.9)

5. Secondary Outcome: Cognitive-Linguistic Quick Test (CLQT)
Description: The following subtests from the CLQT will be administered: Symbol Cancellation, Story Retelling, Generative Naming, Symbol Trails, Design Memory, Mazes,and Design Generation. These scores will be used to calculate composite scores for the cognitive domains of Attention, Executive Function (EF), and Visuospatial skills (VS). Some tests are weighted more than others in each composite score, by multiplying the score as follows and then adding the scores together: Attention = Symbol Cancellation (x9), Story Retelling (x2), Symbol Trails (x3), Mazes (x4), and Design Generation (x1); EF = sum of Symbol Trails, Generative Naming, Mazes, and Design Generation; VS = Symbol Cancellation (x2), Symbol Trails (x2), Design Memory (x4), Mazes (x3), Design Generation (x1). For all composite scores, a low number indicates greater deficit. For Attention, the highest score is 215 and lowest is 0. For EF, the highest score is 40 and lowest is 0. For VS, the highest score is 105 and lowest is 0
Time Frame: Change from baseline to 1 day after treatment
Population: People with aphasia due to left hemisphere stroke
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 23 | 14
scores on a scale
  Attention Composite Score Baseline | 150.0 (46.4) | 175.5 (33.1)
  Attention Composite Score 1 day post-treatment | 155.9 (50.3) | 184.9 (21.2)
  Executive Function Composite Score Baseline | 21.9 (6.5) | 23.7 (5.8)
  Executive Function Composite Score 1 Day Post | 23.1 (7.6) | 25.3 (5.6)
  Visuospatial Function Composite Score Baseline | 78.6 (17.6) | 86.7 (12.9)
  Visuospatial Function Composite Score 1 Day Post | 80.7 (20.4) | 91.4 (12.6)

6. Secondary Outcome: Reading Assessments
Description: A set of reading tasks designed to assess oral reading of real words and non-words at the single word level. The list of real words consisted of 142 words. A score of 0 indicates no words were read correctly and a score of 142 indicates all words were read correctly. The non-word test included 30 non-words. A score of 0 indicates no non-words were read correctly and a score of 30 indicates that all non-words were read correctly.
Time Frame: Change from baseline to 1 day after treatment
Population: People with aphasia due to left hemisphere stroke
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 23 | 14
scores on a scale
  Reading Real Words Baseline | 89.1 (51.2) | 85.1 (61.7)
  Reading Real Words 1 Day Post-treatment | 89.7 (50.5) | 87.3 (59.2)
  Reading Non-words Baseline | 6.1 (6.3) | 8.9 (8.8)
  Reading Non-words 1 Day Post-treatment | 6.3 (7.4) | 8.5 (8.0)

7. Secondary Outcome: Motricity Index
Description: An assessment of upper extremity motor impairment, including: pinch grip, elbow flexion, and shoulder abduction. For pinch grip, which consisted of holding a small plastic cube between the thumb and index finger, scoring was as follows: 0=No movement, 11=Beginnings of prehension, 19=Grips cube but unable to hold against gravity, 22=Grips cube, held against gravity but not against weak pull, 26=Grips cube against pull but weaker than left side, 33=Normal pinch grip. For elbow flexion and shoulder abduction, scoring was as follows: 0=No movement, 9=Palpable contraction in muscle but no movement, 14=Movement seen but not full range/not against gravity, 19=Full range against gravity, not against resistance, 25=Movement against resistance but weaker than left side, 33=Normal power. Both the right and the left side were tested.
Time Frame: Change from baseline to 1 day after treatment
Population: People with aphasia due to left hemisphere stroke
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 23 | 14
scores on a scale
  Pinch Grip Left Baseline | 33 (0) | 33 (0)
  Pinch Grip Left 1 Day Post-treatment | 33 (0) | 33 (0)
  Elbow Flexion Left Baseline | 33 (0) | 33 (0)
  Elbow Flexion Left 1 Day Post-treatment | 33 (0) | 33 (0)
  Shoulder Abduction Left Baseline | 32.6 (1.7) | 33 (0)
  Shoulder Abduction Left 1 Day Post-treatment | 33 (0) | 33 (0)
  Pinch Grip Right Baseline | 25.9 (10.2) | 19.1 (15.9)
  Pinch Grip Right 1 Day Post-treatment | 25.9 (10.3) | 18.4 (16.6)
  Elbow Flexion Right Baseline | 22.4 (12.2) | 19.0 (14.9)
  Elbow Flexion Right 1 Day Post-treatment | 24.0 (11.7) | 19.0 (14.9)
  Shoulder Abduction Right Baseline | 22.9 (11.7) | 17.0 (15.0)
  Shoulder Abduction Right 1 Day Post-treatment | 21.7 (12.7) | 17.4 (14.9)

ADVERSE EVENTS:
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/14
Other Adverse Events (participants affected / at risk) | 0/24 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No